CLINICAL TRIAL: NCT05754983
Title: To Evaluate the Prognostic Risk Factors and Long-term Health Effects of Immunotherapy Patients Based on the Specific Disease Cohort Registered With Patients
Brief Title: Risk Factors and Long-term Impact of ICIs
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSL-020
Record Dates: First submitted 2023-01-10; First posted 2023-03-06 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood sample, cancer tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Solid tumor patients receiving immunotherapy for the first time were included in the study — Solid tumor patients receiving immunotherapy were included in the study. Baseline information before treatment (including demographic characteristics, basic diseases and their medication history, tumor and anti-tumor history, quality of life scores, etc.) and follow-up information after treatment (PFS, OS, etc.) were collected to summarize factors that may affect the efficacy and prognosis of patients receiving immunotherapy

SUMMARY:
This study plans to conduct a multicenter, observable and controlled cohort study to solid-tumor patients with receiving immunotherapy and to collect information about their treatment related efficacy, adverse events and health status to build a disease cohort database based on patient reports, and then analyze the risk factors affecting the efficacy, prognosis and adverse events of immunotherapy and the impact of immunotherapy on health status. It is expected to provide high-level evidence-based medical evidence for the selection of immunotherapy schemes for these patients, the precise prevention and health management of adverse events after immunotherapy, and the further improvement of survival prognosis of patients

DETAILED DESCRIPTION:
This study is intended to conduct a multicenter, observable and controlled cohort study in multiple clinical centers including the First Affiliated Hospital of Xi'an Jiaotong University to solid-tumor patients who received immunotherapy for the first time. The baseline information before treatment was collected (mainly including three collection methods, namely, patients' self filling information, physician assisted filling information, and medical record system import information. The information collected was mainly in the following aspects: demographic characteristics, tumor and anti-tumor information, gene testing information, blood sample collection information, and questionnaire evaluation information) and follow-up information after treatment (The collection method and content are the same as the baseline information.) Collect the relevant factors that may affect the treatment efficacy and prognosis of patients, build a prospective disease cohort database based on patient reports, and then analyze the risk factors that affect the efficacy, prognosis and adverse events of immunotherapy and the impact of immunotherapy on health status. We also retrospectively collected some data from medicine records for validation. The outcome indicators are mainly disease free progression survival (PFS), The secondary indicators were the total survival period (OS), objective response rate (ORR), immune-related adverse events (irAEs) and the scoring results of various questionnaires (PHQ-9, etc). It is expected to provide high-level evidence-based medical evidence for the selection of immunotherapy schemes for these patients, the precise prevention and health management of adverse events after immunotherapy, and the further improvement of survival prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age range of subjects: the age of subjects is no less than 18 years old;
* Receiving any ICIs treatment or ICIs combined with other treatments;
* Soild malignant tumor proved by pathology (histology or cytology);
* First treatment with ICIs {including ICIs (first) combined with other treatments)};
* Any stage and treatment line (new auxiliary, auxiliary and advanced treatment)
* Willing to treat, and can come to the hospital regularly in the later period

Exclusion Criteria:

* Previous medical history of other malignant tumors;
* No pathology (histology or cytology) certificate;
* Having received ICIs or other immunotherapy in the past;
* Participated in clinical research in the past and may have applied ICIs or other immunotherapy;
* Weak treatment intention or long-term treatment in other hospitals/departments

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The included population is malignant solid tumor patients receiving immunotherapy for the first time
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | Two years
  It refers to the time from randomization to disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospitap of Xian Jiaotong University, Xi’an, Shanxi, China